CLINICAL TRIAL: NCT02852811
Title: Reducing Menopausal Symptoms for Women During Menopause Using Group Education in a Primary Health Care Setting: A Randomized Controlled Trial
Brief Title: Reducing Menopausal Symptoms for Women During Menopause Using Group Education in a Primary Health Care Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: fou2016; registration number: 041-09 (Registry Identifier: The Regional Ethical Review Board)
Record Dates: First submitted 2016-05-26; First posted 2016-08-02 (Estimated); Last update posted 2016-08-02 (Estimated); Status verified 2016-05

CONDITIONS: Menopause
Keywords: Climacteric; Education; Mental health; Menopause
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- group education (Other): To measure improvement of menopause symptoms and depression all participating women answered a baseline questionnaire and a follow-up questionnaire four month later. The questionnaires who were used: The Menopause Rating Scale (MRS) and The Montgomery-Asberg Depression Rating Scale (MADRS). MRS were used for reflecting menopause symptom and MADRS for depression symptoms.
  Interventions: Other: Group education
- control group (No Intervention): The control group did not obtain any group education or any other intervention. Women answered at baseline questionnaire and four month later. The questionnaires who were used: The Menopause Rating Scale (MRS) and The Montgomery-Asberg Depression Rating Scale (MADRS). MRS were used for reflecting menopause symptom and MADRS for depression symptoms.

INTERVENTIONS:
Other: Group education — Intervention involving two education session with topics common in menopause transition.
  Arms: group education

SUMMARY:
The aim of the study is to investigate if group education about the topic menopause to women in PHC can improve women's menopausal symptoms and reduce depression.

DETAILED DESCRIPTION:
One hundred twenty women will be included in the study. The survey population consists of Swedish-speaking women aged 45-55 years and seek care at Distriktsköterskemottagningen in Skene and at the Antenatal clinic in Svenljunga. The selection is done consecutively.

Method:

Grouping:The women will be randomly allocated to intervention group and control group (60/60).

The intervention:

The project includes the implementation of a total of four equivalent group treatments. Two of the group education will be at Skene Medical center and two Svenljunga Medical center. Group treatments are carried out by the district nurse and midwife in common. Each treatment group includes 15 women. A total of 60 women will thus participate in group education..Each treatment group consists of two information sessions of 2 hours.

The first information contains information about the menstrual cycle, hormonal shift, urogenital symptoms, and information on prevention and health promotion self-care.

The other information currently contains information about cardiovascular risk factors during menopause, relations, mental health, information about depressive symptoms and for preventive measures and health-promoting self-care.

The control group did not obtain any group education or any other intervention.

ELIGIBILITY:
Inclusion Criteria:

* female gender, 45 to 55 years of age, comprehension and fluency in the Swedish language.

Exclusion Criteria:

* that the patient did not any longer want to participate in the study.

Ages: 45 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 131 (Actual)
Dates: Start 2009-10; Primary Completion 2011-06 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change in menopause symptoms during baseline to four month follow up. The measurement that be used were The Menopause Rating Scale (MRS). | from baseline to four month follow up
  Primary outcome measure: Change in menopausal symptoms (using the menopause rating scale).
Change in depression symptoms during baseline to four month follow up. The measurement that be used was The Montgomery-Asberg Depression Rating Scale (MADRS). | from baseline to four month follow up
  Primary outcome measure: Change in depression score (using the Montgomery-Asberg depression rating scale)

CONTACTS AND LOCATIONS:
Overall Officials: Gun Rembeck, PhD, Principal Investigator — Research and Development Center Södra Älvsborg, Närhälsan, Research and Development, Primary Health Care Region, Västra Götaland, Sweden,

IPD SHARING:
Plan to Share IPD: No